CLINICAL TRIAL: NCT02475954
Title: Telehealth Cognitive-Behavioral Therapy for Depression in Parkinson's Disease
Brief Title: Telehealth Cognitive Behavioral Therapy for Depression in Parkinson's Disease (PD)
Acronym: TH-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Department of Veterans Affairs, New Jersey (U.S. Federal Agency); Rutgers Robert Wood Johnson Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-353
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Depression; Parkinson's Disease
Keywords: Depression; Telehealth; Parkinson's Disease; Veterans; Care-partners; Cognitive-Behavioral Therapy; Caregiver
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TH-CBT + Standard Care (Active Comparator): Cognitive-behavioral therapy delivered via telehealth with a focus on decreasing depressive symptoms in Parkinson's Disease (PD).
  Interventions: Behavioral: TH-CBT; Other: Standard Care
- Standard Care (Other): VA standard care depression in Parkinson's Disease (PD)
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: TH-CBT — The TH-CBT group will receive the study intervention and standard care. The study treatment has been previously manualized and modified for remote administration, as described in the introduction to the revised application.12 PD Veterans will receive 10 weekly individual sessions (60 minutes each) of CBT, delivered via Video-to-Home (V2H).
  Arms: TH-CBT + Standard Care
Other: Standard Care — Standard Care is defined as medical and psychiatric treatment provided by patients' personal doctors (e.g., neurologists, psychiatrists, therapists). Veterans will continue to receive routine clinical care and will remain on all depression treatments that they were receiving prior to their study (e.g., stable anti-depressant medications, established psychotherapy, clinical monitoring).

SUMMARY:
When Veterans with Parkinson's disease (PD) suffer from depression, they are more likely to experience disease complications, interpersonal difficulties with caregivers, and poorer quality of life. Unfortunately, depression in Veterans with PD is inadequately treated at the current time. Treatment for depressed Veterans with PD will require the elimination of geographical barriers to care and approaches that address the unique aspects of PD. The proposed study will be the first to explore a novel and innovative, PD-informed psychotherapy package for depressed Veterans with PD and their Caregivers, delivered through video-to-home telehealth. If the results of this proposal are promising, a much needed treatment can be made available to Veterans with PD and their Caregivers across the country, regardless of geographical location.

DETAILED DESCRIPTION:
Objective: There is a critical need for treatments that address depression and barriers to mental health care among the nearly 100,000 Veterans with Parkinson's Disease (PD) served by the VA. Depression in PD (dPD) is a major complicating factor in the movement disorder, affecting several key functional outcomes such as motor disability, cognitive status, quality of life, and caregiving relationships. The challenge to meeting the treatment needs of Veterans with dPD centers on the lack of clinicians who are knowledgeable about the interactions of PD and depression, the considerable transportation barriers faced by this population, combined with the geographical dispersion of specialized services within the VA, and the paucity of effectiveness research that informs treatments for dPD. The proposed study seeks to overcome these challenges by using a telehealth delivery platform (i.e., video-to-home) to test the effectiveness of a 10-session cognitive-behavioral treatment (CBT) package that has been tailored to address the unique needs of depressed Veterans with PD. The proposed treatment package also provides support and skills-training to the Veteran's Caregiver (3 sessions). This HSR&D proposal will be the first to: 1) to evaluate the effectiveness of TH-CBT for improving Veteran outcomes in dPD, 2) to examine the impact of TH-CBT for dPD on a variety of Caregiver outcomes, and 3) to assess Veteran and Caregiver perspectives on TH-CBT using a mixed-methods sequential explanatory design.

Method: A PD-informed, telehealth-administered cognitive behavioral therapy package (TH-CBT) for dPD will be evaluated in a clinical effectiveness trial. 180 participants (90 Veterans and 90 Caregivers) will be enrolled. Half of the sample will receive the study treatment package (TH-CBT), in addition to their standard medical care. The other half will only receive standard medical care. The two groups will be compared at baseline, midpoint (week 5), endpoint (week 10), and 1 and 6 months post treatment. Veterans will be assessed with standard measures of depression, anxiety, quality of life, and motor function, while Caregivers will be evaluated with measures of caregiver burden, empowerment, and communication.

Impact: Given the public health impact of improved depression treatment in Veterans with Parkinson's disease, the knowledge to be gained may be significant and the project could directly impact clinical practice. The data gleaned from this study will guide the wide-scale implementation of this remote care model within the VA for meeting the specialized needs of Veterans with PD. Towards this goal, successful results for the proposed study will facilitate a multisite initiative to further examine issues of dissemination, implementation, and effectiveness, using a hybrid research design. Ultimately, these Health Science Research & Development (HSR&D) data may support the development of a centralized care model, in which highly specialized dPD providers, concentrated in a few locations, provide specialty care to Veterans and Caregivers across the country.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PD diagnosis in the VA medical record
* Primary Major Depression, Dysthymia, or Depression Not Otherwise Specified (NOS) of at least moderate severity per the Structured Clinical Interview (SCID) for Diagnostic and Statistical Manual of Mental Disorders (DSM5) Disorders.
* Access to a computer/tablet with high-speed internet access. primary
* Ages 35-85
* Stable medication and mental health regimen greater than or equal to 6 weeks, including:

  * applicable antidepressants
  * other psychotropic agents
  * movement disorder drugs
  * clinic-based psychotherapies
* Willingness to involve a family member or friend to participate

Exclusion Criteria:

* Possible dementia or marked cognitive impairment [Montreal Cognitive
* Assessment Score (MoCA) less than 21
* Motor fluctuations greater than or equal to 50% of the day
* Suicidal plans or intent (determined by clinical interview)
* Unstable medical conditions

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Interian, PhD, Principal Investigator — Lyons Campus of the VA New Jersey Health Care System, Lyons, NJ
Locations (1):
- Lyons Campus of the VA New Jersey Health Care System, Lyons, NJ, Lyons, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pontone GM, Dissanayaka N, Dobkin RD, Mari L, Marsh L, Vernaleo BA, Weintraub D, Mari Z. Integration and Extension of Specialty Mental Healthcare Services to Community Practice in Parkinson Disease. Am J Geriatr Psychiatry. 2019 Jul;27(7):712-719. doi: 10.1016/j.jagp.2019.03.005. Epub 2019 Mar 13. PMID 30955991
- [Result] Dobkin RD, Mann SL, Weintraub D, Rodriguez KM, Miller RB, St Hill L, King A, Gara MA, Interian A. Innovating Parkinson's Care: A Randomized Controlled Trial of Telemedicine Depression Treatment. Mov Disord. 2021 Nov;36(11):2549-2558. doi: 10.1002/mds.28548. Epub 2021 Mar 12. PMID 33710659

RESULTS

PARTICIPANT FLOW:
Groups:
- TH-CBT + Standard Care: Cognitive-behavioral therapy delivered via telehealth with a focus on decreasing depressive symptoms in Parkinson's Disease (PD).
  TH-CBT: The TH-CBT group will receive the study intervention and standard care. The study treatment has been previously manualized and modified for remote administration, as described in the introduction to the revised application.12 PD Veterans will receive 10 weekly individual sessions (60 minutes each) of CBT, delivered via Video-to-Home.
  Standard Care: Standard Care is defined as medical and psychiatric treatment provided by patients' personal doctors (e.g., neurologists, psychiatrists, therapists). Veterans will continue to receive routine clinical care and will remain on all depression treatments that they were receiving prior to their study (e.g., stable antidepressant medication, established psychotherapy, clinical monitoring).
Period: Overall Study
Arm/Group | TH-CBT + Standard Care | Standard Care
Started | 87 | 87
Completed | 73 | 75
Not Completed | 14 | 12
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 11 | 9
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard Care: VA standard care depression in Parkinson's Disease (PD)
  Standard Care: Standard Care is defined as medical and psychiatric treatment provided by patients' personal doctors (e.g., neurologists, psychiatrists, therapists). Veterans will continue to receive routine clinical care and will remain on all depression treatments that they were receiving prior to their study (e.g., stable antidepressant medication, established psychotherapy, clinical monitoring).
- Total: Total of all reporting groups
Arm/Group | TH-CBT + Standard Care | Standard Care | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.27 (7.79) | 66.42 (9.51) | 66.84 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One person had missing data.
  Participants
    number analyzed (Participants) | 87 | 86 | 173
    Female | 41 | 39 | 80
    Male | 46 | 47 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 82 | 86 | 168
    Hispanic or Latino | 7 | 4 | 11
    Not Hispanic or Latino | 75 | 82 | 157
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 84 | 85 | 169
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 4 | 10
    White | 75 | 80 | 155
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Scale Scores: Min:0 and Max: 52. Higher scores mean a worse outcome. Population: Hamilton Depression Rating Scale was only given to veterans not care partners.
  units on a scale
    number analyzed (Participants) | 45 | 45 | 90
    (all) | 21.60 (4.30) | 22.49 (3.85) | 22.04 (4.08)
Hamilton Anxiety Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale Scores: Min:0 and Max: 56. Higher scores mean a worse outcome. Population: Hamilton Anxiety Rating Scale was only given to veterans, not care partners.
  units on a scale
    number analyzed (Participants) | 45 | 45 | 90
    (all) | 23.49 (4.57) | 24.16 (4.14) | 23.82 (4.35)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment Scores: Min:0 and Max: 30. Higher scores mean a better outcome. Population: This assessment was only given to veterans not care partners.
  units on a scale
    number analyzed (Participants) | 45 | 45 | 90
    (all) | 25.17 (2.72) | 25.00 (2.43) | 25.08 (2.57)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale
Description: This measure uses the Hamilton Depression Rating Scale (HDRS) to express the average severity of depressive symptoms, with higher scores indicating greater depression. Hamilton Depression Rating Scale (HAMD) Score Min:0 and Max: 52. Higher scores mean a worse outcome.
Time Frame: 10 weeks (endpoint) and 6 months post-treatment
Population: This assessment was only given to veterans not care partners.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TH-CBT + Standard Care | Standard Care
Number analyzed (Participants) | 45 | 45
score on a scale
  10 weeks (endpoint) | 16.46 (5.18) | 21.37 (5.27)
  6 months post-treatment | 16.35 (4.97) | 20.70 (5.47)

2. Other Pre Specified Outcome: Family Empowerment Scale
Description: The Family Empowerment scale measures the degree to which caregivers feel empowered to help care for their Veteran. To obtain a score for each area, sum the item responses where "Not at all" is scoring as 1, "Mostly not true" is scored as 2, "Somewhat true" is scored as 3, "Mostly true" is scored as 4, and "Very true" is scored as 5 to produce a score ranging from 12-60. The items are scored in the same direction, i.e., no item scores are reversed, and a higher score indicates relatively more empowerment in each respective area. Higher scores mean a better outcome.
Time Frame: 10 weeks (endpoint) and 6 months post-treatment
Population: This assessment was only given to care partners not veterans. Some care partners did not complete the Family Empowerment Scale at 6-months post treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TH-CBT + Standard Care | Standard Care
Number analyzed (Participants) | 44 | 43
score on a scale
  10 weeks (endpoint) | 49.82 (6.20) | 44.06 (9.12)
  6 months post-treatment: number analyzed (Participants) | 39 | 40
  6 months post-treatment | 49.66 (7.47) | 45.31 (7.04)

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | TH-CBT + Standard Care | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/87 | 1/87
Serious Adverse Events (participants affected / at risk) | 9/87 | 12/87
Other Adverse Events (participants affected / at risk) | 9/87 | 9/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-CBT + Standard Care (N=87) | Standard Care (N=87)
Cardiac related (Cardiac disorders) | 3 (3) | 1 (1)
Endocrine related (Endocrine disorders) | 1 (1) | 0 (0)
GI related (Gastrointestinal disorders) | 0 (0) | 2 (2)
General disorders related (General disorders) | 0 (0) | 1 (1)
Infection related (Infections and infestations) | 0 (0) | 2 (2)
Nervous system related (Nervous system disorders) | 4 (4) | 1 (1)
Renal related (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscle related (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-CBT + Standard Care (N=87) | Standard Care (N=87)
Muscle related (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Cancer related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Nervous system related (Nervous system disorders) | 4 (4) | 2 (2)
Cardiac related (Cardiac disorders) | 0 (0) | 1 (1)
GI related (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary related (Renal and urinary disorders) | 0 (0) | 1 (1)
General disorders related (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study has several limitations that merit comment. This sample was 100% male, which may limit the generalizability of findings to females. In order to provide direct policy guidance on the additive value of V-CBT to VA's current standard of PD care, we utilized an existing-practice control (TAU). It is not possible to fully disaggregate effects of this V-CBT intervention from nonspecific factors (e.g., therapeutic relationship, attention) that contribute to all psychotherapy outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02475954/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02475954/ICF_001.pdf